CLINICAL TRIAL: NCT05326958
Title: Repeatability of Static & Dynamic Composite Confocal Microscopy for Assessment of the Corneal Nerve Fiber Plexus in Early Diabetic Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: E-2015-1
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Normal Eyes of Subjects Without Diabetes Mellitus; Subjects With Diabetes Mellitus Type 2 Without Coexisting DPN; Subjects With Diabetes Mellitus Type 2 With Coexisting Early to Moderate DPN

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Eyes of Subjects without DM (Experimental): Study Part 1 conducted at only site 1 . Single measurement made on 3 separate visits at site 1 (total 3 images acquired) with HRT RCM and HRT RCM-E functional module (investigational).
  Interventions: Device: HRT RCM; Device: HRT RCM-E
- Eyes of DM Type 2 subjects without coexisting DPN (Experimental): Study part 2 conducted at site 2.
  1 image acquired with HRT RCM-E functional module (investigational).
  Interventions: Device: HRT RCM-E
- Eyes of DM Type 2 subjects with coexisting early to moderate DPN (Experimental): Study part 2 conducted at site 2.
  1 image acquired with HRT RCM-E functional module (investigational).
  Interventions: Device: HRT RCM-E

INTERVENTIONS:
Device: HRT RCM — Imaging with HRT RCM done only at site 1 (on normal eyes of subjects without DM).
  Other Names: Heidelberg Engineering Retina Tomograph HRT 3 with the Rostock Cornea Module (HRT RCM)
  Arms: Normal Eyes of Subjects without DM
Device: HRT RCM-E — imaging done on eyes of all enrolled subjects at site 1 and site 2.
  Other Names: Heidelberg Engineering Retina Tomograph HRT 3 with the Rostock Cornea Module EyeGuidance functional module (HRT RCM-E)

SUMMARY:
This prospective study was was divided into 2 parts and carried out at 2 sites in Germany.

Part 1 assessed Repeatability in healthy, non-diabetic population (Group "control").

Part 2 collected data to evaluate the diagnostic and prognostic value of using Heidelberg Engineering Retina Tomograph (HRT) 3 with the Rostock Cornea Module EyeGuidance functional module (HRT RCM-E) in subjects with early to moderate DPN (Groups"none" and "mild", respectively).

DETAILED DESCRIPTION:
Part 1 aimed to evaluate the diagnostic and prognostic value of the optimized dynamic composite corneal nerve plexus image acquisitions done with HRT RCM-E compared to standard static composite image acquisition with Heidelberg Engineering Retina Tomograph (HRT) 3 with the Rostock Cornea Module (HRT RCM).

The part 2 (research part) evaluated changes in corneal nerve plexus parameters in diabetes patients without or with early to moderate Diabetic Peripheral Neuropathy (DPN) and correlated the observed changes with progression of early DPN.

ELIGIBILITY:
Inclusion Criteria:

* All

  * Able and willing to undergo the test procedures, give consent, and to follow instructions.
  * Signed informed consent.
  * ≥18 years.
* Part 1, Site 1

  * Normal eyes of patients without Diabetes Mellitus
  * Fasting blood glucose < 100 mg/dl
  * HbA1c ≤ 6.5%
* Part 2, Site 2

  * Diabetes Mellitus Type 2 without coexisting DPN (NSS score ≤2 and / or NDS score ≤2)
  * Diabetes Mellitus Type 2 with coexisting early to moderate DPN. (NSS score 3-4 and / or NDS score 3-5)
  * 6.5% < HbA1c ≤ 9.5%

Exclusion Criteria:

* Vulnerable subjects (Such as: individuals with lack of or loss of autonomy due to immaturity or through mental disability, persons in nursing homes, children, impoverished persons, subjects in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Other vulnerable subjects include, for example, members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel (if linked to CI site), employees of the sponsor, members of the armed forces (if linked to CI site or sponsor), and persons kept in detention.)
* Subjects unable to read or write
* Contact lens wearers (soft and rigid)
* Patients with symptomatic dry eye
* Patients with conjunctivitis at the time of inclusion
* Patients with history of corneal surgery
* Patients with diabetic retinopathy
* Patients with history of neuronal diseases that according to the expertise of the investigator might have an influence on corneal nerve fiber plexus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
corneal nerve fiber length (CNFL) | Through study completion, an average of 1 day to upto 3 days
  Acquired image processed to obtain parameters required to calculate nerve fibre metrics
corneal nerve fiber density (CNFD) | Through study completion, an average of 1 day to upto 3 days
  Acquired image processed to obtain parameters required to calculate nerve fibre metrics
average corneal nerve single fiber length (CNSFL) | Through study completion, an average of 1 day to upto 3 days
  Acquired image processed to obtain parameters required to calculate nerve fibre metrics
average weighted corneal nerve fiber tortuosity (CNFTo) | Through study completion, an average of 1 day to upto 3 days
  Acquired image processed to obtain parameters required to calculate nerve fibre metrics
corneal nerve branch density (CNBD) | Through study completion, an average of 1 day to upto 3 days
  Acquired image processed to obtain parameters required to calculate nerve fibre metrics
corneal nerve connecting points (CNCP) | Through study completion, an average of 1 day to upto 3 days
  Acquired image processed to obtain parameters required to calculate nerve fibre metrics
average weighted corneal nerve fiber thickness (CNFTh) | Through study completion, an average of 1 day to upto 3 days
  Acquired image processed to obtain parameters required to calculate nerve fibre metrics

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Rudolf Guthoff, Principal Investigator — Universitätsmedizin Rostock; Univ.Prof.Dr.med.Dr.h.c.Diethelm Tschöpe, Principal Investigator — Herz- und Diabeteszentrum NRW, UKRUB, Universitätsklinik der Ruhr Universität Bochum; Priv.-Dozent Dr. med.Hans-Joachim Hettlich — Augen-Praxisklinik Minden

REFERENCES:
- [Derived] Matuszewska-Iwanicka A, Stratmann B, Stachs O, Allgeier S, Bartschat A, Winter K, Guthoff R, Tschoepe D, Hettlich HJ. Mosaic vs. Single Image Analysis with Confocal Microscopy of the Corneal Nerve Plexus for Diagnosis of Early Diabetic Peripheral Neuropathy. Ophthalmol Ther. 2022 Dec;11(6):2211-2223. doi: 10.1007/s40123-022-00574-z. Epub 2022 Oct 3. PMID 36184730